CLINICAL TRIAL: NCT03343860
Title: Is Ablation of All Inducible Atrial Tachycardias an Appropriate Endpoint During Redo Procedures After Initial Persistent AF Ablation? A Multi-center, Randomised, Single-blind Study
Brief Title: Catheter Ablation of All Inducible AT Post AF Ablation
Acronym: INDUCATH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AZ Sint-Jan AV (Other)
Responsible Party: Principal Investigator, Sebastien Knecht, Professor Doctor, AZ Sint-Jan AV
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2097
Record Dates: First submitted 2017-11-08; First posted 2017-11-17 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Atrial Tachycardia; Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional (Active Comparator): PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. Inducibility will be tested but no ablation will be carried out and a DCC post AT mapping will be performed if necessary. The procedure will end up after these steps.
  Interventions: Procedure: AT case 1.1; Procedure: AT case 1.2; Procedure: AT case 1.3; Procedure: AT case 1.4; Procedure: SR Case 1
- Non inducibility (Active Comparator): PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. Then inducibility will be tested and all inducible AT will be mapped and ablated (max 5 consecutive AT) .
  Interventions: Procedure: AT case 2.1; Procedure: AT case 2.2; Procedure: AT case 2.3; Procedure: AT case 2.4; Procedure: SR Case 2

INTERVENTIONS:
Procedure: AT case 1.1 — In the case of AT at the time of ablation :
  In the case of sinus rhythm restoration, PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. Inducibility will be tested but no ablation will be carried out and a DCC post AT mapping will be performed if necessary. The procedure will end up after these steps.
  Arms: Conventional
Procedure: AT case 2.1 — In the case of AT at the time of ablation :
  In the case of sinus rhythm restoration, PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. Then inducibility will be tested and all inducible AT will be mapped and ablated (max 5 consecutive AT)
  Arms: Non inducibility
Procedure: AT case 1.2 — In the case of AT at the time of ablation :
  In the case of termination to another AT, a DCC will be performed. Thereafter, PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. Inducibility will be tested but no ablation will be carried out and a DCC post AT mapping will be performed if necessary. The procedure will end up after these steps.
  Arms: Conventional
Procedure: AT case 1.3 — In the case of AT at the time of ablation :
  In the case of AF deterioration, a DCC will be performed. Thereafter, PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. Inducibility will be tested but no ablation will be carried out and a DCC post AT mapping will be performed if necessary. The procedure will end up after these steps
  Arms: Conventional
Procedure: AT case 1.4 — In the case of AT at the time of ablation :
  In the case of no AT termination, a DCC will be performed. Thereafter, PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. Inducibility will be tested but no ablation will be carried out and a DCC post AT mapping will be performed if necessary. The procedure will end up after these steps.
  Arms: Conventional
Procedure: AT case 2.2 — In the case of AT at the time of ablation :
  In the case of termination to another AT, ablation of the subsequent AT will be performed until sinus rhythm restoration. Thereafter, PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. Then inducibility will be tested and all inducible AT will be mapped and ablated (max 5 consecutive AT)
  Arms: Non inducibility
Procedure: AT case 2.3 — In the case of AT at the time of ablation :
  In the case of AF deterioration, a DCC will be performed. Thereafter, PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. Then inducibility will be tested and all inducible AT will be mapped and ablated (max 5 consecutive AT)
  Arms: Non inducibility
Procedure: AT case 2.4 — In the case of AT at the time of ablation :
  In the case of no AT termination, a DCC will be performed. Thereafter, PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. Then inducibility will be tested and all inducible AT will be mapped and ablated (max 5 consecutive AT)
  Arms: Non inducibility
Procedure: SR Case 1 — In the case of SR at the time of ablation:
  PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. The CTI line will be performed in all patients with a ECG showing a typical counterclockwise flutter. Inducibility will be tested but no ablation will be carried out and a DCC post AT mapping will be performed if necessary. The procedure will end up after these steps.
  Arms: Conventional
Procedure: SR Case 2 — In the case of SR at the time of ablation:
  PV will be re-isolated if necessary and lines (CTI, roof and mitral) already blocked during the first procedure will be re-blocked if necessary. The CTI line will be performed in all patients with a ECG showing a typical counterclockwise flutter. Then inducibility will be tested and all inducible AT will be mapped and ablated (max 10 consecutive AT)
  Arms: Non inducibility

SUMMARY:
In the treatment of symptomatic drug resistant persistent atrial fibrillation (Ps AF), catheter ablation has a class IIA indication. During the follow-up, a significant amount of patients (~50%) will experience atrial tachycardias (AT) recurrence. The endpoint of AT ablation during the second procedure has not been validated. At present, several strategies are considered as good clinical practice.

Main objective: To evaluate if ablation of all inducible AT post AF ablation (ATPAFA) offers as substantial benefit in comparison with ablation of the clinical ATPAF only during a redo procedure post initial persistent AF ablation.

Secondary objectives:

To evaluate the prognosis of non-inducibility during a redo procedure for ATPAFA

ELIGIBILITY:
Inclusion Criteria:

* Male or Female Adults (≥18 years old)
* Patients with stable ATPAF at least two months after the first AF ablation procedure.
* Consent signed by the patient after reading the information leaflet

Exclusion Criteria:

* Mental or physical inability to take part in the study
* Spontaneous AF in the EP lab
* Presence of any pulmonary vein stents
* Presence of any pre-existing pulmonary vein stenosis
* Presence of any cardiac valve prosthesis
* Clinically significant mitral valve regurgitation or stenosis
* Myocardial infarction, PCI / PTCA or coronary artery stenting within the last 3 months
* Unstable angina
* Any cardiac surgery within the last 3 months
* NYHA class III or IV congestive heart failure
* Uncontrolled hyperthyroidism

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2017-04-05 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Freedom from any documented episode of AT or AF lasting longer than 30 seconds without AAD and occurring during the 1 year follow-up after the ATPAF ablation procedure. | During 12 months follow-up
  There will be a 1-months blanking period after ATPAF ablation. A repeated left atrial ablation at any time (even during the blanking period) will be considered as a recurrence.

SECONDARY OUTCOMES:
The number of non-inducible ATPAFA during a redo procedure | At repeat procedure(s) during the 12 months follow-up
Incidence of repeat procedures | During 12 months follow-up
Incidence of procedure related complications | During 12 months follow-up
Procedure time | Baseline
Fluoroscopy duration | Baseline
Correlation of the AT mechanism during the redo procedure with the AT Mechanism during the index procedure | At repeat procedure(s) during the 12 months follow-up
  To evaluate the correlation between the ATPAFA mechanism during the index procedure with potential AT mechanism during the follow up (in the case of AT recurrence)

CONTACTS AND LOCATIONS:
Overall Officials: Sebastien Knecht, MD, PhD, Principal Investigator — sebastien.knecht@azsintjan.be
Locations (6):
- Department Clinical Trial Cardiology, Bruges, Belgium
- France (2):
  - Hôpital Cardiologique d Haut Leveque, Bordeaux
  - CHU Toulouse, Toulouse
- Germany (2):
  - Medizinische Klinik und Poliklinik, Universitätsmedizin Mainz, Mainz
  - Deutsches Herzzentrum München, Munich
- St Thomas Hospital London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided